CLINICAL TRIAL: NCT03045848
Title: Prospective Multicenter Observational Study for Evaluating Efficacy and Safety of Biofreedom Stent in Patients With Coronary Artery Disease (Biofreedom Registry)
Brief Title: Biofreedom Prospective Multicenter Observational Registry
Status: Terminated | Type: Observational
Why Stopped: Impossible device delivery because of sponsor change
Sponsor: Wonju Severance Christian Hospital (Other)
Collaborators: Cordis US Corp. (Industry)
Responsible Party: Principal Investigator, Junghan Yoon, Professor, Wonju Severance Christian Hospital
Other Study IDs: Biofreedom V2.2
Record Dates: First submitted 2017-01-29; First posted 2017-02-08 (Estimated); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Coronary Artery Disease Aggravated; Myocardial Ischemia; Myocardial Infarction
Keywords: Observational registry; All-comers open label registry; Drug coated stent; Multicenter; Stenting; Coronary Artery Disease; Coronary revascularization; Percutaneous Coronary Intervention
MeSH Terms: conditions — Myocardial Ischemia; Myocardial Infarction; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Biofreedom drug-coated stent: Subject implanted Biofreedom DCS for coronary artery disease
  Interventions: Device: Biofreedom drug-coated stent

INTERVENTIONS:
Device: Biofreedom drug-coated stent — BioFreedom (Biosensors International Technologies, Singapore) is the only polymer- and carrier-free drug coated stent with Biolimus A9 in a selectively micro-structured abluminal surface. It is a stainless steel bare metal surface with 120 micron thick corrugated ring strut.

SUMMARY:
LEADERS-FREE trial demonstrated the safety and efficacy of polymer-free drug-coated stent (Biofreedom, Biosensors International Technologies, Singapore) in patients with high bleeding risk. But, there are limited clinical evidences for extending these findings to generalized patients who are eligible to PCI. Therefore, the purpose of this registry is to evaluate the safety and efficacy of Biofreedom stent in patients with coronary artery disease.

DETAILED DESCRIPTION:
Percutaneous coronary intervention (PCI) and related interventional cardiology field are rapidly growing in current era. First generation drug eluting stent (DES) needed long-term dual antiplatelet therapy (DAPT) for preventing future stent thrombosis. But, second generation DES showed better clinical outcomes in terms of target lesion revascularization and stent thrombosis. Later, polymer technology that was used to release drugs gradually improved. BASKET-PROVE II trial compared biodegradable polymer (BP) DES (Nobori, Terumo) with durable polymer DES (Xience Prime, Abbott Vascular) and bare metal stent (ProKinetik, Biotronik) for the safety and efficacy in 2-year follow-up. BP-DES showed 7.6% of event rates in composite endpoint including cardiac death, myocardial infarction (MI), clinically indicated target-vessel revascularization (TVR) which was non-inferior to DP-DES(6.8%) and superior to bare metal stent (12.7%). There were no statistical differences for the event rates of stent thrombosis, MI and cardiac death among three groups in 1-year follow-up. Biodegradable polymer has begun to emerge and suggested the possibility of shortening the duration of DAPT. LEEDERS-FREE trial was designed to confirm the safety and efficacy of polymer-free drug-coated stent (Biofreedom, Biosensors International Technologies, Singapore) compared to bare metal stent (Gazelle stent, Biosensors International Technologies, Singapore) in patients with high bleeding risk. During 390 days, drug coated stent showed significant superiority to bare metal stent for the safety composite endpoint (cardiac death, MI or stent thrombosis) (9.4% vs. 12.9%, P=0.0005). Clinically-driven target-lesion revascularization also showed significant differences between drug-coated stent (5.1%) and bare metal stent (9.8%) (P<0.001). This results provided new therapeutic options that DAPT duration could be shortened to 1 month in patients with high bleeding risk. The rate of cardiovascular events was relatively higher than second generation DES. However, this result should be carefully interpreted because the main purpose of LEADERS-FREE trial is to enroll high bleeding risk patients who are generally excluded in second generation DES studies. Additional studies are needed because there are limited clinical evidences for extending these findings of LEADERS-FREE trial to generalized patients who are eligible to PCI.

ELIGIBILITY:
Inclusion Criteria:

* Subject with ≥ 19 years
* Subject implanted with Biofreedom DCS within 1 month
* Subject who decided to participation and signed informed consent

Exclusion Criteria:

* Known intolerance to heparin, aspirin, clopidogrel, biolimus, cobalt chromium or contrast media (Subject with hypersensitivity to contrast media controlled by steroid and pheniramine can be included this study, but subject with anaphylaxis to contrast media will be excluded).
* Pregnancy
* Woman who have a plan of pregnancy during study period
* Subject with life expectancy less than 12 months
* Subject with cardiogenic shock
* Subject treated with other drug-eluting stent (DES), bioresorbable vascular scaffold (BVS) or bare metal stent (BMS)
* Subject participating in other randomized controlled study with DES, BVS or BMS

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All-comers patient population with all subjects requiring coronary revascularization with a drug-coated stent (DCS)
Sampling Method: Non-Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
Device-oriented composite end point (TLF) | 12 months
  Composite of cardiac death, any myocardial infarction not clearly attributable to a nontarget vessel, and clinically indicated target-lesion revascularization

SECONDARY OUTCOMES:
Patient-oriented composite end point | 12 months
  Composite of any death, any myocardial infarction, and any revascularization
Cardiac death | 12 months
Non-cardiac death | 12 months
Any myocardial infarction | 12 months
Any myocardial infarction not clearly attributable to a non-target vessel | 12 months
Any revascularization | 12 months
Clinically indicated target-lesion revascularization | 12 months
Clinically indicated target-vessel revascularization | 12 months
ARC defined stent thrombosis | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Junghan Yoon, MD, PhD, Study Director — Yonsei University
Locations (16):
- South Korea (16):
  - Dankook University Hospital, Cheonan, Chungcheongnam-do
  - Kangwon National University School of Medicine, Chuncheon, Gangwon-do
  - Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Soonchunhyang University Bucheon Hospital, Bucheon-si, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon, Gyeonggi-do
  - CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Yeungnam University Medical Center, Daegu, Gyeongsangbuk-do
  - Daegu Catholic University Medical Center, Daegu, Gyeongsangbuk-do
  - Pusan National University Yangsan Hospital, Pusan, Gyeongsangnam-do
  - Eulji General Hospital, Seoul
  - KyungHee University at Gangdong, Seoul
  - Gangnam Severance Hospital, Seoul
  - Chung-Ang University Hospital, Seoul
  - Seoul National University Boramae Medical Center, Seoul
  - Veterans Health Service Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Undecided